CLINICAL TRIAL: NCT02262156
Title: Treatment Of Depression In Patients With Temporal Lobe Epilepsy: Comparative Study Of Cognitive Behavioral Therapy Vs. Selective Serotonin Reuptake Inhibitors
Brief Title: CBT Versus Selective Serotonin Reuptake Inhibitor For Treatment Of Depression In Temporal Lobe Epilepsy Patients
Acronym: CBTvsSSRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Edgar Daniel Crail Melendez, Md, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49/06; U1111-1158-3147 (Other: WHO UTN)
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-10

CONDITIONS: Depression; Epilepsy, Temporal Lobe
Keywords: Cognitive Behavioral Therapy; Selective serotonin reuptake inhibitor; depression; epilepsy
MeSH Terms: conditions — Depression; Epilepsy, Temporal Lobe; Epilepsy | interventions — Cognitive Behavioral Therapy; Selective Serotonin Reuptake Inhibitors; Antidepressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral Therapy (Experimental): CBT program to be used in group modality that focused on managing symptoms of depression in patients with epilepsy.
  12 CBT sessions, consisting of one weekly 90-minute session for 12 consecutive weeks.
  Interventions: Other: Cognitive behavioral therapy
- Selective serotonin euptake inhibitor (Active Comparator): Patients will receive a SSRI (sertraline or citalopram) for 12 weeks. Dose will be adjusted every 4 weeks according to medical criteria.
  Interventions: Drug: SSRI

INTERVENTIONS:
Other: Cognitive behavioral therapy — The CBT group will receive 12 weekly 90-minute sessions. Each session will be given in group form by one certified CBT therapist and one neuropsychiatrist in training on group therapy.
  The CBT structure include psychoeducation, addressing dysfunctional thoughts and maladaptive behaviors; problem solving techniques, assertiveness, coping strategies and depression relapse prevention
  Other Names: CBT
  Arms: Cognitive behavioral Therapy
Drug: SSRI — Patients will receive the "treatment as usual" with a SSRI: sertraline or citalopram. In patients already taking antidepressants for more than 8 weeks before enrollment but still experiencing depressive symptoms, treatment could be optimized either by augmenting the dose of his antidepressant or by changing to one of the SSRI mentioned.
  Other Names: selective serotonin reuptake inhibitor; antidepressant
  Arms: Selective serotonin euptake inhibitor

SUMMARY:
The aim of the study is to compare the effect of group-cognitive-behavioral therapy (CBT)versus treatment as usual with the selective serotonin reuptake inhibitor sertraline, in patients with diagnosis of temporal lobe epilepsy (TLE) and depressive disorder.

DETAILED DESCRIPTION:
patients with temporal lobe epilepsy and depression will be enrolled into one of two treatment modality. The first group will receive 12 group cognitive behavioral sessions. CBT is a psychotherapy focused on the recognition and change of distorted thoughts and maladaptive behaviors.

The second group will receive treatment with the selective serotonin reuptake inhibitor sertraline or citalopram for 12 weeks. This antidepressant is wide used to treat depression in patients with TLE.

ELIGIBILITY:
Inclusion Criteria:

* With Major depressive disorder according to criteria from the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* Diagnosed with TLE according to the criteria of the International League Against Epilepsy
* Literates had sign an informed consent
* Patients on antidepressant treatments will be allowed to participate only if they had been at stable doses for more than 8 weeks and still show signs of significant depression

Exclusion Criteria:

* Patients with high risk of suicide who required hospitalization
* Patients who abused or are dependent on drugs
* Those with a history of head trauma six months prior to the interview
* Patients who have any condition that would prevent them from understanding the study or the psychotherapeutic process, such as mental retardation, psychosis, delirium, dementia, etc
* Patients who have previously received CBT
* Patients who have started, an antidepressant drug the last 8 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory score | baseline, 6 weeks and 12 weeks

SECONDARY OUTCOMES:
Quality of Life in Epilepsy Scale | baseline, 6 weeks and 12 weeks
  the quality of life in epilepsy scale measures the patients perceived quality of life. Higher score indicates better quality of life. score goes from 0 to 100
Hospital anxiety and depression scale (HADS) | baseline, 4weeks and 12 weeks
  the HADS measures severity of symptoms of anxiety and depression. Lower scores indicates less symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crail-Melendez, MD, Principal Investigator — El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía MVS, México, D.f., Mexico

REFERENCES:
- [Derived] Maguire MJ, Marson AG, Nevitt SJ. Antidepressants for people with epilepsy and depression. Cochrane Database Syst Rev. 2021 Apr 16;4(4):CD010682. doi: 10.1002/14651858.CD010682.pub3. PMID 33860531